CLINICAL TRIAL: NCT04273594
Title: BLOC: Prospective, Multi-Center, Study of Subjects Undergoing FemBloc Permanent Contraception With Two Confirmation Procedures (FemBloc With FemChec and Fluoro HSG)
Brief Title: FemBloc® Permanent Contraception - Confirmation Feasibility Trial
Acronym: BLOC
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Femasys Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CP-100-008
Record Dates: First submitted 2020-02-14; First posted 2020-02-18 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Contraception
Keywords: permanent contraception; birth control; pregnancy prevention

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- FemBloc (Experimental): Investigational device and procedure
  Interventions: Device: FemBloc

INTERVENTIONS:
Device: FemBloc — Treatment with FemBloc for women who desire permanent birth control (female sterilization)

SUMMARY:
The trial objectives include evaluating the adequacy of proposed mitigations for the previous pivotal trial of the FemBloc Permanent Contraceptive System and validating the confirmation procedure by comparing FemChec (ultrasound) to fluoroscopic hysterosalpingogram (fluoro HSG) for post-occlusion in the same patient.

ELIGIBILITY:
Inclusion Criteria:

* Female, 21 - 45 years of age desiring permanent birth control
* Sexually active with male partner
* Regular menstrual cycle for last 3 months or on hormonal contraceptives

Exclusion Criteria:

* Uncertainty about the desire to end fertility
* Known or suspected pregnancy
* Prior tubal surgery, including sterilization attempt
* Prior endometrial ablation
* Presence, suspicion, or previous history of gynecologic malignancy
* Abnormal uterine bleeding requiring evaluation or treatment
* Scheduled to undergo concomitant intrauterine procedures at the time of procedure(s)
* Allergy to shellfish, betadine or iodinated contrast

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Reliance Rate | within 1 year
  Number of subjects told to rely divided by number of qualified subjects
Concordance | within 1 year
  Concordance between FemBloc confirmation with FemChec and Fluoro HSG confirmation

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - New Horizons Clinical Trials, Chandler, Arizona
  - Precision Trials AZ, LLC, Phoenix, Arizona
  - Midtown OB GYN North, Columbus, Georgia
  - Women's Health Advantage, Fort Wayne, Indiana
  - Saginaw Valley Medical Research Group, Saginaw, Michigan
  - University Hospitals - Cleveland Medical Center, Beachwood, Ohio